CLINICAL TRIAL: NCT00029263
Title: R-21 Project: Screening Herbs for Drug Interference
Brief Title: Screening Herbs for Drug Interactions
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: R21AT000511-01 (NIH)
Record Dates: First submitted 2002-01-09; First posted 2002-01-10 (Estimated); Last update posted 2006-08-18 (Estimated); Status verified 2006-07

CONDITIONS: Healthy

INTERVENTIONS:
Drug: herbals

SUMMARY:
The purpose of this study is to detect potential herb-drug interactions in volunteers.

DETAILED DESCRIPTION:
The use of herbal medicines in the treatment of various medical and psychiatric conditions has accelerated in the last decade. It has also become evident that herbal medications are being used concomitantly with conventional prescription and over-the-counter medications. However, the systematic evaluation of the potential of these agents to interact with conventional medications has been generally neglected. Compounding this problem is the fact that even single entity herbal products can contain a multitude of naturally occurring chemicals which serve as candidates for potential herb-drug interactions by inhibiting or inducing specific hepatic isozymes. Numerous reports document the importance of pharmacokinetic interactions involving inhibition or induction of the cytochrome P450 (CYP) enzyme system. In this study, the ten most commonly used herbal products in the US will be systematically evaluated for inhibition of CYP 3A4 and 2136, and induction of CYP 3A4. Collectively, these enzyme systems are involved in the metabolism of approximately 80% of all marketed medications.

Participants in this study will receive a single dose of the prescription drug alprazolam and the over-the-counter cough suppressant, dextromethorphan on two occasions. A combination of probe drugs will be given to normal volunteers both in the absence and presence of herbal medications. The plasma and urine concentration of these agents and their respective metabolites will be determined in order to evaluate individual herbal products degree and specificity of enzyme inhibitory or inductive effects.

ELIGIBILITY:
Inclusion Criteria:

* Normal healthy volunteers who are taking no medications.
* Must be non-smokers.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140
Dates: Start 2001-08; Study Completion 2004-05

CONTACTS AND LOCATIONS:
Overall Officials: John Markowitz, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Institute of Psychiatry, Medical University of SC, Charleston, South Carolina, United States